CLINICAL TRIAL: NCT06352593
Title: Role of Intraoperative Dexmedetomidine Infusion in Endovascular Intervention for Aneurysmal Subarachnoid Hemorrhage: A Randomized Controlled Trial
Brief Title: Intraoperative Dexmedetomidine Infusion in Endovascular Intervention for Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36264PR557/2/24
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Dexmedetomidine; Infusion; Endovascular; Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Dexmedetomidine) (Experimental): Patients will be administered Dexmedetomidine 0.5 μg/kg for 10 min and then 0.4 μg/kg/h adjusted to 0.2-0.6 μg/kg/h.
  Interventions: Drug: Intraoperative Dexmedetomidine
- Group C (placebo group) (Placebo Comparator): Patients will receive normal saline (control group) .
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intraoperative Dexmedetomidine — Patients will be administered DEX 0.5 μg/kg for 10 min and then 0.4 μg/kg/h adjusted to 0.2-0.6 μg/kg/h.
  Arms: Group D (Dexmedetomidine)
Other: Placebo — Patients will receive normal saline.
  Arms: Group C (placebo group)

SUMMARY:
The aim of this study is to evaluate the role of intraoperative dexmedetomidine infusion in endovascular intervention for aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage is a sudden, life-threatening emergency caused by bleeding in the subarachnoid space between the brain and skull. Cerebral vasospasm (VSP) is the leading risk factor of neurological deterioration (i.e., delayed cerebral ischemia [DCI] and cerebral infarction) after aneurysmal subarachnoid hemorrhage (SAH) and a cause of morbidity and mortality.

Dexmedetomidine (DEX) is a highly selective α-2 adrenergic receptor agonist. The α -2 receptor agonists have a long track record of use for sedation and analgesia. It has been shown that α -2 agonists are neuroprotective in craniocerebral and subarachnoid injuries. Dexmedetomidine has a significant effect on the central nervous system and decreases the blood flow in the brain and the requirement or needs for cerebral oxygen. It also modifies memory and enhances cognitive ability effects like sedation, analgesic, and anxiolytics. Dexmedetomidine is shown to decrease catecholamine in the brain and improves the perfusion ability in the penumbra. The glutamate level is significantly reduced by Dexmedetomidine (DEX), and so injuries at the cellular level is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) I-III
* Unruptured subarachnoid hemorrhage (SAH) confirmed by digital subtraction catheter angiography (DSA) undergoing endovascular intervention with general anesthesia.

Exclusion Criteria:

* Subarachnoid hemorrhage (SAH) from a lesion other than a ruptured saccular aneurysm.
* Intraventricular or intracerebral blood in the absence of localized thick or diffuse Subarachnoid hemorrhage (SAH).
* No or localized thin subarachnoid hemorrhage (SAH) on computed tomography (CT).
* Cerebral vasospasm on admission digital subtraction catheter angiography (DSA).
* Hypotension (systolic blood pressure 90 mm Hg) refractory to fluid therapy.
* Neurogenic pulmonary edema.
* Cardiac failure requiring inotropic support.
* Severe or unstable concomitant condition or disease or chronic condition.
* Kidney and/or liver disease.
* Prior cerebral damage on computed tomography (CT) scan such as stroke (>2 cm maximum diameter).
* Pregnancy.
* Traumatic brain injury.
* Previously treated cerebral aneurysm.
* Arterial venous malformation.
* Pre-existing cerebrovascular disorder that will affect diagnosis and evaluation of Subarachnoid hemorrhage (SAH).
* Ischemic heart disease or second or third-degree atrioventricular block.
* Long-term abuse of alcohol, opioids, or sedative-hypnotic drugs.
* Obesity (body mass index [BMI] >30 kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-04-06 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Incidence of vasospasm | 14 days after intervention
  Vasospasm is quantified as the percent reduction in arterial diameter between baseline and digital subtraction catheter angiography (DSA). A global assessment of vasospasm will then made and classified as none/mild (0% to 33%), moderate (34% to 66%), or severe (67% to 100%).

SECONDARY OUTCOMES:
Incidence of morbidity and mortality (M/M) | 6 weeks after intervention
  Morbidity and mortality (M/M) is defined as at least one of the following: death within 6 weeks of subarachnoid hemorrhage (SAH) from any cause; new cerebral infarct within 6 weeks of subarachnoid hemorrhage(SAH) compared with post-procedure computed tomography (CT) scan; delayed ischemic neurological deficit (DIND) due to vasospasm within 14 days of subarachnoid hemorrhage (SAH); and rescue therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author